CLINICAL TRIAL: NCT00343135
Title: An Open, Non-comparative Study to Evaluate the Efficacy and Safety of AUGMENTIN 1gm (875mg Amoxicillin/125mg Clavulanic Acid) po q 12 Hours in the Treatment of Uncomplicated Skin and Soft Tissue Infections in Pakistan
Brief Title: AUGMENTIN 1gm In Skin And Soft Tissue Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103997
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Skin Diseases, Infectious; Infection, Soft Tissue
Keywords: Skin; AUGMENTIN; 1gm; Soft; tissue; Infections
MeSH Terms: conditions — Skin Diseases, Infectious; Soft Tissue Infections; Infections | interventions — Amoxicillin

ARMS (1):
- ARM 1 (Experimental)
  Interventions: Drug: amoxicillin/clavulanate potassium 1gm

INTERVENTIONS:
Drug: amoxicillin/clavulanate potassium 1gm — amoxicillin/clavulanate potassium 1gm

SUMMARY:
Study to evaluate the effects of AUGMENTIN 1gm in the treatment of Skin and Soft tissue infections

ELIGIBILITY:
Inclusion Criteria:

* having diagnosed uncomplicated soft tissue infection (e.g furuncle, cellulitis)
* has given freely documented consent.

Exclusion Criteria:

* antibiotics
* have renal or hepatic insufficiency
* systemic toxicity
* pregnancy
* lactation
* hypersensitivity to penicillin or Beta-lactam antibiotics

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2004-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Clinical response at 10 - 14 days post therapy | 10 - 14 days

SECONDARY OUTCOMES:
Clinical response at on-therapy evaluation visit (2 - 4 days following initiation of therapy and 48 - 96 hours post therapy) Bacteriological response at (2 - 4 days following initiation of therapy, 48 - 96 hours post therapy, 10 - 14 days post therapy) | 2 - 4 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Pakistan (2):
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore